CLINICAL TRIAL: NCT04083625
Title: the Effect of Carbetocin in Decreasing Intraoperative Blood Loss in Abdominal Myomectomy: a Randomized Controlled Trial
Brief Title: the Effect of Carbetocin in Decreasing Intraoperative Blood Loss in Abdominal Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Myomectomy uterotonic
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Abdominal Myomectomy
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbetocin (Experimental): 100microgram in 10 cm syringe carbetocin IV just before skin incision of myomectomy.
  Interventions: Drug: carbetocin 100 mcg
- placebo (Placebo Comparator): 10 cm syringe normal saline IV given just before skin incision of myomectomy.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: carbetocin 100 mcg — a 10 cm syringe containing 100 mcg carbetocin just before skin incision of myomectomy.
  Arms: carbetocin
Drug: placebo — a 10 cm syringe normal saline IV given just before skin incision of myomectomy.
  Arms: placebo

SUMMARY:
To investigate the effectiveness of carbetocin on reducing intraoperative blood loss during abdominal myomectomy

ELIGIBILITY:
Inclusion Criteria:

* • Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging

  * Age ≥ 25 years and ≤ 50 years
  * Pre-operative hemoglobin >10 g/dl
  * Ability to understand and the willingness to sign a written informed consent.
  * Admissible medical/surgical history
  * Five or less symptomatic uterine myomas
  * symptomatic stage 3 to 6 fibroids, according to FIGO staging

Exclusion Criteria:

* • Post-menopausal women

  * Patients with known bleeding/clotting disorders
  * Patients with a history of gynecologic malignancy
  * Hypertension.
  * Cardiac and Pulmonary diseases.
  * History of allergic reactions attributed to carbetocin

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Mean amount of intraoperative blood loss | intraoperative
  Mean amount of intraoperative blood loss in ml

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University
Locations (1):
- Giza hospital, Giza, Egypt

REFERENCES:
- [Derived] Taher A, Farouk D, Mohamed Kotb MM, Ghamry NK, Kholaif K, A Mageed A Allah A, Ali AS, Osman OM, Nabil H, Islam Y, Bakry MS, Islam BA, Alalfy M, Nassar SA, Bosilah AH, Ghanem AA, Ali Rund NM, Refaat R, Abdel Wahed Ali HA, Bakry A, Ashour ASA, Nabil M, Zaki SS. Evaluating efficacy of intravenous carbetocin in reducing blood loss during abdominal myomectomy: a randomized controlled trial. Fertil Steril. 2021 Mar;115(3):793-801. doi: 10.1016/j.fertnstert.2020.09.132. Epub 2021 Jan 16. PMID 33461754